CLINICAL TRIAL: NCT03046316
Title: Local Consolidative Therapy (LCT) in Patients With Advanced Stage Non-small Cell Lung Cancer Who do Not Progress After Front Line Systemic Therapy
Brief Title: Local Therapy in Advanced NSCLC With Non-progressive Disease (PD) After First Line Therapy
Acronym: LOCAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Dr., Guangdong Association of Clinical Trials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1602
Record Dates: First submitted 2016-11-29; First posted 2017-02-08 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Lung Neoplasms
Keywords: Therapeutics; local therapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- local consolidative treatment (Other): Patients will be referred to multiple disciplinary treatment discussion for the decision of local consolidative treatment to primary or metastatic lesions including surgery, radiotherapy or interventional therapy.
  Interventions: Other: local consolidative treatment

INTERVENTIONS:
Other: local consolidative treatment — local consolidative treatment to primary or metastases, which includes surgery, radiotherapy or interventional therapy

SUMMARY:
This is a prospective single arme real-world study clinical study, which aims to investigate the overall benefit and safety of consolidative therapy in advanced NSCLC (stage III/IV) patients , who do not progress after front line systemic therapy (chemotherapy, target therapy or immunological checkpoint inhibitors).

DETAILED DESCRIPTION:
It is required that pathological diagnosis and genetic profile including epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK) and ROS proto-oncogene 1 (ROS1) be established prior to enrollment. Standard front line systemic should be given according to clinical practice. Molecular targeting drugs for patients with driving mutations should be acquired legally. Patients without driving mutations should undergo standard first line chemotherapy and or immunological checkpoint inhibitors. One cycle is three weeks and response evaluation is done every two cycles. CR, PR and SD should be confirmed after four cycles of therapy.

Patients, who achieve non-PD after four cycles of treatment, with distant metastasis involving no more than five total metastatic lesions, will be screened and enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age >= 18 years, with life expectancy of at least 12 weeks.
* Patients with histologically documented metastatic (stage IV) non-small cell lung cancer.
* Subjected to driving genes examination including EGFR, ALK and ROS1.
* Achieve complete response (CR)/partial response (PR)/stable disease (SD) after front line systemic treatment (chemotherapy, targeted therapy or immunological checkpoint inhibitors).
* Total metastatic lesions is limited to five.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of <= 2.
* Patients must have measurable disease according to the RECIST (version 1.1) criteria.
* Adequate organ function as defined by the following criteria:

  * Liver function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 upper limit of normal (ULN) in the absence of liver metastases or up to 5 ULN in case of liver metastases. Total bilirubin <= 1.5 ULN.
  * Bone marrow function: Granulocyte count >= 1,500/mm3 and platelet count ≥100,000/mm3 and hemoglobin >= 80g/dl.
  * Renal function: serum creatinine <= 1.5 ULN or creatinine clearance >= 60 ml/min. (based on modified Cockcroft-Gault formula).
  * Adequate coagulating function.
* For all females of childbearing potential a negative serum/urine pregnancy test must be obtained within 48 hours before enrollment. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Males must agree to use effective contraception during the study period and for at least 12 weeks after completion of the study treatment.
* Written (signed) informed Consent to participate in the study.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Stage I-III a NSCLC completing radical treatment , then undergoing systemic anti-cancer treatment after recurrence.
* Patients with PFS no more than 3 months. to first line theray.
* Patients with history of any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).
* Prior palliative surgery or other local therapy specifically directed against advanced lung cancer.
* Contraindication for localized treatment including surgery, radiotherapy or interventional therapy judged by physicians.
* Patients with any unstable systemic disease (including active infections, significant cardiovascular disease, any significant hepatic, renal or metabolic disease).
* Patients who are at risk (in the investigator's opinion) of transmitting human immunodeficiency virus (HIV) through blood or other body fluids.
* Nursing or lactating women.
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
* Patients who has mental disorder or other disease that contribute to no compliance.
* Unwilling to write informed consent to participate in the study.
* Patients who is unwilling to accept the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 8 months
  month

SECONDARY OUTCOMES:
Response rate | 6 months
  percentage(%)
Lung Cancer Symptom Scale | 12 months
  quality of life
overall survival | 2 years
  month

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Guangdong General Hospital&Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong General Hospital, Guangzhou, Guagndong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barlesi F, Scherpereel A, Rittmeyer A, Pazzola A, Ferrer Tur N, Kim JH, Ahn MJ, Aerts JG, Gorbunova V, Vikstrom A, Wong EK, Perez-Moreno P, Mitchell L, Groen HJ. Randomized phase III trial of maintenance bevacizumab with or without pemetrexed after first-line induction with bevacizumab, cisplatin, and pemetrexed in advanced nonsquamous non-small-cell lung cancer: AVAPERL (MO22089). J Clin Oncol. 2013 Aug 20;31(24):3004-11. doi: 10.1200/JCO.2012.42.3749. Epub 2013 Jul 8. PMID 23835708
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Suzuki H, Yoshino I. Approach for oligometastasis in non-small cell lung cancer. Gen Thorac Cardiovasc Surg. 2016 Apr;64(4):192-6. doi: 10.1007/s11748-016-0630-7. Epub 2016 Feb 19. PMID 26895202
- [Background] Shimada Y, Saji H, Kakihana M, Kajiwara N, Ohira T, Ikeda N. Survival outcomes for oligometastasis in resected non-small cell lung cancer. Asian Cardiovasc Thorac Ann. 2015 Oct;23(8):937-44. doi: 10.1177/0218492315596463. Epub 2015 Jul 22. PMID 26207006
- [Background] Pan H, Simpson DR, Mell LK, Mundt AJ, Lawson JD. A survey of stereotactic body radiotherapy use in the United States. Cancer. 2011 Oct 1;117(19):4566-72. doi: 10.1002/cncr.26067. Epub 2011 Mar 15. PMID 21412761
- [Background] Rusthoven KE, Kavanagh BD, Cardenes H, Stieber VW, Burri SH, Feigenberg SJ, Chidel MA, Pugh TJ, Franklin W, Kane M, Gaspar LE, Schefter TE. Multi-institutional phase I/II trial of stereotactic body radiation therapy for liver metastases. J Clin Oncol. 2009 Apr 1;27(10):1572-8. doi: 10.1200/JCO.2008.19.6329. Epub 2009 Mar 2. PMID 19255321
- [Background] Rusthoven KE, Kavanagh BD, Burri SH, Chen C, Cardenes H, Chidel MA, Pugh TJ, Kane M, Gaspar LE, Schefter TE. Multi-institutional phase I/II trial of stereotactic body radiation therapy for lung metastases. J Clin Oncol. 2009 Apr 1;27(10):1579-84. doi: 10.1200/JCO.2008.19.6386. Epub 2009 Mar 2. PMID 19255320
- [Background] Wronski M, Arbit E, Burt M, Galicich JH. Survival after surgical treatment of brain metastases from lung cancer: a follow-up study of 231 patients treated between 1976 and 1991. J Neurosurg. 1995 Oct;83(4):605-16. doi: 10.3171/jns.1995.83.4.0605. PMID 7674008
- [Background] Nakagawa H, Miyawaki Y, Fujita T, Kubo S, Tokiyoshi K, Tsuruzono K, Kodama K, Higashiyama M, Doi O, Hayakawa T. Surgical treatment of brain metastases of lung cancer: retrospective analysis of 89 cases. J Neurol Neurosurg Psychiatry. 1994 Aug;57(8):950-6. doi: 10.1136/jnnp.57.8.950. PMID 8057119
- [Background] Jett JR, Schild SE, Kesler KA, Kalemkerian GP. Treatment of small cell lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e400S-e419S. doi: 10.1378/chest.12-2363. PMID 23649448
- [Background] Patel AN, Simone CB 2nd, Jabbour SK. Risk factors and management of oligometastatic non-small cell lung cancer. Ther Adv Respir Dis. 2016 Aug;10(4):338-48. doi: 10.1177/1753465816642636. Epub 2016 Apr 8. PMID 27060187
- [Background] Barone M, Di Nuzzo D, Cipollone G, Camplese P, Mucilli F. Oligometastatic non-small cell lung cancer (NSCLC): adrenal metastases. Experience in a single institution. Updates Surg. 2015 Dec;67(4):383-7. doi: 10.1007/s13304-015-0336-x. Epub 2015 Nov 20. PMID 26589602
- [Background] Raz DJ, Lanuti M, Gaissert HC, Wright CD, Mathisen DJ, Wain JC. Outcomes of patients with isolated adrenal metastasis from non-small cell lung carcinoma. Ann Thorac Surg. 2011 Nov;92(5):1788-92; discussion 1793. doi: 10.1016/j.athoracsur.2011.05.116. Epub 2011 Sep 22. PMID 21944257
- [Background] DeLuzio MR, Moores C, Dhamija A, Wang Z, Cha C, Boffa DJ, Detterbeck FC, Kim AW. Resection of oligometastatic lung cancer to the pancreas may yield a survival benefit in select patients--a systematic review. Pancreatology. 2015 Sep-Oct;15(5):456-462. doi: 10.1016/j.pan.2015.03.014. Epub 2015 Apr 3. PMID 25900320
- [Background] Lencioni R, Crocetti L, Cioni R, Suh R, Glenn D, Regge D, Helmberger T, Gillams AR, Frilling A, Ambrogi M, Bartolozzi C, Mussi A. Response to radiofrequency ablation of pulmonary tumours: a prospective, intention-to-treat, multicentre clinical trial (the RAPTURE study). Lancet Oncol. 2008 Jul;9(7):621-8. doi: 10.1016/S1470-2045(08)70155-4. Epub 2008 Jun 17. PMID 18565793
- [Derived] Dong S, Wang Z, Zhang JT, Yan B, Zhang C, Gao X, Sun H, Li YS, Yan HH, Tu HY, Liu SM, Gong Y, Gao W, Huang J, Liao RQ, Lin JT, Ke EE, Xu Z, Zhang X, Xia X, Li AN, Liu SY, Pan Y, Yang JJ, Zhong WZ, Yi X, Zhou Q, Yang XN, Wu YL. Circulating Tumor DNA-Guided De-Escalation Targeted Therapy for Advanced Non-Small Cell Lung Cancer: A Nonrandomized Controlled Trial. JAMA Oncol. 2024 Jul 1;10(7):932-940. doi: 10.1001/jamaoncol.2024.1779. PMID 38869865